CLINICAL TRIAL: NCT03720106
Title: The Way to Goal-oriented Therapy Planning in Neurorehabilitation: Adherence to Targeted Clinical Pathways in Subacute Stroke- a Feasibility Study
Brief Title: The Way to Goal-oriented Therapy Planning in Neurorehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehaklinik Zihlschlacht AG (Other)
Collaborators: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RZS_01_2018
Record Dates: First submitted 2018-10-04; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Stroke Rehabilitation; Triage
Keywords: interdisciplinarity; therapy planning; assessment; stroke; neurorehabilitation; physical therapy; occupational therapy; neuropsychology; logopedia
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Other): In this arm the GOAL therapy plan is used.
  Interventions: Other: GOAL therapy plan

INTERVENTIONS:
Other: GOAL therapy plan — The GOAL algorithm designs a therapy plan based on the LIMOS assessment, patient goals and subject-specific treatment pathways. The adherence of this therapy plan is examined.

SUMMARY:
The aim of this feasibility study is to investigate whether target-oriented treatment planning can be maintained in the rehabilitation of stroke patients using the existing classification (LIMOS) and evidence-based specialist treatment pathways. If the goal-oriented treatment planning cannot be adhered to, reasons for failure should be investigated.

DETAILED DESCRIPTION:
According to Feigin and employees, in 2013 there were 25.7 million people worldwide who survived a stroke. In order to regain independence in everyday life after a mild to severe stroke, a rehabilitation phase is recommended. Rehabilitation is a holistic process with the aim of maximising participation in the daily life of the affected person. Tailor-made interventions with a focus on impairment, activity and participation should be carried out for this purpose. The International Classification of Functioning, Disability and Health (ICF) was developed in a worldwide consensus and declared by the WHO as a generally accepted framework for describing function and health. In rehabilitation, it is considered as standard and is used to speak a uniform language between the disciplines, to understand the needs of patients, to adapt the corresponding interventions to the needs and to measure outcomes. In order to optimally plan the process, Stroke Guidelines recommend to define goals together with the patient and to use standardized and valid assessments. So far, the following assessments have been used for the neurorehabilitation of stroke patients: Barthel Index, Functional Independence Measure and Functional Assessment Measure as well as the Modified Ranking Scale, but according to Ottiger and her colleagues there was a lack of multidisciplinary assessments with good psychometric properties and which are based on ICF. For this reason, the ICF-based multidisciplinary observation scale (LIMOS) was developed in Lucerne. It consists of four multidisciplinary components based on the following ICF domains: motor function, cognition, communication and coping with everyday life. Due to its good psychometric properties, LIMOS was recommended as a multidisciplinary assessment for neurorehabilitation. The Rehabilitation Clinic Zihlschlacht (RZS) has an interprofessional team. Each discipline carries out subject-specific assessments and plans the necessary therapy units based on empirical values. So far, however, there has been no algorithm that records the deficits of a stroke patient on an interdisciplinary basis and uses the results to determine the main therapeutic areas. In RZS, patient satisfaction with the therapy plan in 2017 was 77%. The reasons for dissatisfaction were: Lack of inclusion of needs, lack of adaptation to changing needs, time aspects, lack of information and the proportion of cognitive and motor therapies. Now the therapy planning system is to be optimized. The LIMOS classification should help to record the patient in an interdisciplinary manner and to visualize focal points. Together with the patient, goals are discussed which are weighted on the basis of LIMOS. These results, together with evidence-based subject-specific treatment pathways, are integrated into an algorithm (GOAL) that creates a goal-oriented treatment plan.

The aim of this feasibility study is to investigate whether target-oriented treatment planning can be maintained in the rehabilitation of stroke patients using the existing classification and evidence-based specialist treatment pathways. If the goal-oriented treatment planning cannot be adhered to, reasons for failure should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ischemic (e.g., anterior, middle or posterior cerebral artery, cerebellar arteries) or haemorrhagic stroke
* subacute stage: 2 weeks to 6 months after the event7
* signed declaration of consent

Exclusion Criteria:

* other cerebrovascular events (sinus vein thrombosis or subarachnoid haemorrhage)
* participation in other intervention studies
* any medical conditions that interfere with the patient's ability to adhere to the target therapy plan as judged by the sponsor-investigator (e.g., severe dementia)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity | up to 6 months
  The deviations of the targeted therapy plan are checked weekly on Sunday by the sponsor-investigator. The deviations are documented in %. If there are some deviations, the reasons for the deviations are checked and analysed descriptively.

SECONDARY OUTCOMES:
Patient satisfaction: questionnaire of the RZS | 72 hours before discharge of the patient
  The patient satisfaction is examined using the questionnaire of the RZS. The results are documented descriptively. the questionnaire contains possible answers to a 5-point likertscale. 1: excellent, 2: very good, 3: good, 4: less good, 5: bad or 1: yes, 2: predominant, 3: partial, 4: rather no, 5: no
Therapist satisfaction: PSSUQ | 72 hours before discharge of the patient
  Using the post-study usability questionnaire (PSSUQ), the therapist satisfaction is evaluated and described descriptively. The rating scale includes a 7-point likert scale with 1: strongly applicable and 7: strongly inapplicable.

OTHER OUTCOMES:
Achievement of longterm goals | 72 hours after admission and 72 hours before discharge of the patient
  The long-term goals are defined 72 hours after admission and are evaluated 72 hours before discharge of the patient.
  . The results are dichotomous (1: achieved and 2: not achieved). An overall score in percent is calculated.
Achievement of the overall rehabilitation goals | 72 hours after admission and 72 hours before discharge of the patient
  The rehabilitation goals are defined within the first week 72 hours after admission in the first rehabilitation meeting and evaluated 72h before discharge according to the national measurement plan of the ANQ. The scale is dichotomous (1: achieved and 2: not achieved). An overall score is calculated in %. The results of the primary outcome "Fidelity" are used to examine possible correlations with the results of the goal achievement (long-term goals and rehab goals). The value 1 stands for a strong correlation, while the value 0 stands for no correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tanner, Principal Investigator — Rehaklinik Zihlschlacht
Locations (1):
- Rehaklinik Zihlschlacht, Center for Neurological Rehabilitation, Zihlschlacht, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feigin VL, Norrving B, George MG, Foltz JL, Roth GA, Mensah GA. Prevention of stroke: a strategic global imperative. Nat Rev Neurol. 2016 Sep;12(9):501-12. doi: 10.1038/nrneurol.2016.107. Epub 2016 Jul 22. PMID 27448185
- [Background] Cieza A, Ewert T, Ustun TB, Chatterji S, Kostanjsek N, Stucki G. Development of ICF Core Sets for patients with chronic conditions. J Rehabil Med. 2004 Jul;(44 Suppl):9-11. doi: 10.1080/16501960410015353. PMID 15370742
- [Background] Weimar C, Kurth T, Kraywinkel K, Wagner M, Busse O, Haberl RL, Diener HC; German Stroke Data Bank Collaborators. Assessment of functioning and disability after ischemic stroke. Stroke. 2002 Aug;33(8):2053-9. doi: 10.1161/01.str.0000022808.21776.bf. PMID 12154262
- [Background] Ottiger B, Vanbellingen T, Gabriel C, Huberle E, Koenig-Bruhin M, Pflugshaupt T, Bohlhalter S, Nyffeler T. Validation of the new Lucerne ICF based Multidisciplinary Observation Scale (LIMOS) for stroke patients. PLoS One. 2015 Jun 25;10(6):e0130925. doi: 10.1371/journal.pone.0130925. eCollection 2015. PMID 26110769